CLINICAL TRIAL: NCT02593500
Title: A Single Center, Single Dose, Open-label, Randomized, Two Period Crossover Study to Determine the Bioequivalence of Two Inhalation Formulations Containing Budesonide 200 µg Administered as 3 Puffs (Total Dose of 600 µg) in at Least 52 Healthy Males and Females Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Inhalation Formulations Containing Budesonide 200 µg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reig Jofre Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BUD01
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2014-04

CONDITIONS: Allergy
Keywords: Bioequivalence, budesonide,
MeSH Terms: conditions — Hypersensitivity | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmictan+Test (Treatment Sequence AB) (Experimental): Treatment period 1:
  Budesonide 200 µg (Budesonida Pulmictan® 200 µg: reference product (A)). Pressurized inhalation suspension. Single dose of 600 µg (3 puffs)per treatment period under fasting conditions.
  Treatment period 2:
  Budesonide 200 µg (test product (B)). Pressurized inhalation suspension. Single dose of 600 µg (3 puffs) per treatment period under fasting conditions.
  Interventions: Drug: Budesonida Pulmictan® 200 µg; Drug: Budesonide 200 µg
- Test+Pulmictan (treatment sequence BA) (Experimental): Treatment period 1:
  Budesonide 200 µg (test product (B)). Pressurized inhalation suspension. Single dose of 600 µg (3 puffs) under fasting conditions.
  Treatment period 2:
  Budesonide 200 µg (Budesonida Pulmictan® 200 µg: reference product (A)). Pressurized inhalation suspension. Single dose of 600 µg (3 puffs) under fasting conditions.
  Interventions: Drug: Budesonida Pulmictan® 200 µg; Drug: Budesonide 200 µg

INTERVENTIONS:
Drug: Budesonida Pulmictan® 200 µg
  Other Names: Budesonide 200 µg (reference product (A)).
Drug: Budesonide 200 µg
  Other Names: Budesonide 200 µg (test product (B))

SUMMARY:
A SINGLE CENTER, SINGLE DOSE, OPEN-LABEL, RANDOMIZED, TWO PERIOD CROSSOVER STUDY TO DETERMINE THE BIOEQUIVALENCE OF TWO INHALATION FORMULATIONS CONTAINING BUDESONIDE 200 µg ADMINISTERED AS 3 PUFFS (TOTAL DOSE OF 600 µg) IN AT LEAST 52 HEALTHY MALES AND FEMALES UNDER FASTING CONDITIONS

The study objective is to determine whether the inhaled test product, budesonide 200 µg (pressurized inhalation suspension) and the inhaled reference product, Budesonida Pulmictan® 200 µg (budesonide; pressurized inhalation suspension) are bioequivalent.

For this purpose the PK profile of budesonide will be compared after administration of a single dose of 600 µg (3 puffs) of each of the two inhalation formulations, under fasting conditions.

DETAILED DESCRIPTION:
The sponsor has developed a new formulation (test product) of an existing medication (reference product) which is intended for a variation in the existing marketing authorization.

The proposed study in healthy males and females is designed to establish a PK profile under fasting conditions for the orally inhaled test and reference products to evaluate bioequivalence.

This will be a single-dose, open-label, laboratory-blind, randomized, two-period crossover study with inhalation administered budesonide200 µg conductedunder fasting conditions inat least 52 healthy males and femalesat a single study center.

The study will comprise:

* Screening period, including serum cortisol levels and documented inhalation training, of maximum 21 days;
* Two treatment periods (each of which will include a profile period of 24 hours)separated by a wash-out period of 7 calendar days (minimum number of days based on half-life of the analyte) to 14 calendar days (maximum number of days based on logistical arrangements) between consecutive administrations of the IMP;
* A post-study visit within 72 hours of completion of the last treatment period of the study.

Participants will be assigned randomly to treatment sequence, prior to the first administration of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, 18 years and older (inclusive).
2. Body Mass Index (BMI) between 18.5 and 30 kg/m2 (inclusive).
3. Body mass not less than 50 kg.
4. Medical history,vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigationsmust be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless theinvestigator considers the deviation to be irrelevant for the purpose of the study.
5. Non-smokers or past-smokers who stopped at least 3 months before entering the study.
6. Serum cortisol value ≥ 275 nmol/L.
7. Forced expiratory volume in 1 second (FEV1) ≥ 80% of the predicted value regarding age, height, gender and ethnicity (European Community for Coal and Steel [ECCS]/European Respiratory Society [ERS]).
8. Females, if:

   • Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal, Note: In postmenopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.

   OR

   • Of childbearing potential, the following conditions are to be met: Negative pregnancy test If this test is positive, the participant will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the participant received IMP, every attempt must be made to follow her to term.

   Not lactating Abstaining from sexual activity(if this is the usual lifestyle of the participant) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study Examples of reliable methods of contraception include non-hormonal intrauterine deviceand barrier methods combined with an additional contraceptive method.

   In this study the concomitant use of hormonal contraceptives as well as (cytochrome P450 [CYP] isoenzyme 3A4 [CYP3A4]) inhibitors is NOT allowed within 28 days before the first dosing and throughout the study.

   Other methods, if considered by the investigator as reliable, will be accepted.
9. Written consent given for participation in the study.

Exclusion Criteria:

1. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
2. Current alcohol use > 21 units of alcohol (1 unit of beer = 340 mL, 1 unit of wine = 200 mL and 1 spirits = 25 mL) per week for males and > 14 units of alcohol per week for females.
3. Regular exposure to substances of abuse (other than alcohol) within the past year.
4. Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks prior to the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator.
5. In this study the concomitant use of hormonal contraceptives as well as (cytochrome P450 [CYP] isoenzyme 3A4 [CYP3A4]) inhibitors is NOT allowed within 28 days before the first dosing and throughout the study.
6. Participation in another study with an experimental drug, where the last administrationof the previous IMP was within 8 weeks before the first administration of IMP in this study.
7. Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
8. A major illness during the 3 months before commencement of the screening period.
9. History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
10. Hypersensitivity to lactose, galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption.
11. History of bronchial asthma or any other bronchospastic disease.
12. History of epilepsy.
13. History of porphyria.
14. Current cataracts present.
15. Glaucoma.
16. History of or current candida of mouth.
17. Hypokalemia.
18. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
19. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
20. Diagnosis of hypotension made during the screening period.
21. Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
22. Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
23. Positive testing for human immunodeficiency virus (HIV), Hepatitis B and Hepatitis C.
24. Positive urine screen for drugs of abuse.
25. Positive urine screen for tobacco use.
26. Positive pregnancy test.
27. Unable to demonstrate proper inhalation techniques involved in using the inhalation devices during the screening training session.
28. Immunization using a live organism vaccine within 4 weeks prior to the first dosing of IMP.
29. Any specific investigational product safety concern.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 24 hours
  Maximum observed plasma concentration (Cmax) obtained directly from the concentration-time data
AUC(0-t) | Up to 24 hours
  Area under the plasma concentration versus time curve (AUC), from time zero to t, where t is the time of the last quantifiable concentration (AUC(0-t)).

SECONDARY OUTCOMES:
tmax | Up to 24 hours
  Time to maximum observed plasma concentration (tmax).
AUC (0-infinity) | Up to 24 hours
  Area under the plasma concentration versus time curve (AUC), with extrapolation to infinity (AUC(0-infinity)).
Terminal elimination rate constant (λz) | Up to 24 hours
Apparent terminal elimination half-life (t1/2). | Up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, Bloemfontein, South Africa